CLINICAL TRIAL: NCT04003376
Title: Efficacy of Fractional CO2 Laser Alone and as Transepidermal Drug Delivery for Different Modalities of Treatment in Alopecia Areata
Brief Title: Efficacy of Fractional CO2 Laser as a Mono- or Adjuvant Therapy for Alopecia Areata
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A Ghazally, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO2LASERAA
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Alopecia Areata
Keywords: fractional carbon dioxide laser
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- fractional carbon dioxide laser alone (Active Comparator): six sessions of fractional carbon dioxide laser will be done for 10 patients with alopecia areata
  Interventions: Device: fractional carbon dioxide laser alone
- fractional carbon dioxide laser and triamcinolone acetonide (Experimental): six sessions of fractional carbon dioxide laser will be done for 10 patients with alopecia areata followed immediately by topical application of triamcinolone acetonide (10mg/ml)
  Interventions: Device: fractional carbon dioxide laser alone; Drug: Triamcinolone Acetonide 10mg/mL
- fractional carbon dioxide laser and platelet rich plasma (Experimental): six sessions of fractional carbon dioxide laser will be done for 10 patients with alopecia areata followed immediately by topical application of autologous platelet rich plasma
  Interventions: Device: fractional carbon dioxide laser alone; Biological: platelet rich plasma
- fractional carbon dioxide laser and vitamin D solution (Experimental): six sessions of fractional carbon dioxide laser will be done for 10 patients with alopecia areata followed immediately by topical application of vitamin D solution
  Interventions: Device: fractional carbon dioxide laser alone; Drug: vitamin D solution

INTERVENTIONS:
Device: fractional carbon dioxide laser alone — six sessions of fractional carbon dioxide laser will be done for alopecia areata lesions
Drug: Triamcinolone Acetonide 10mg/mL — six sessions of fractional carbon dioxide laser will be done for 10 patients with alopecia areata followed immediately by topical application of triamcinolone acetonide
  Arms: fractional carbon dioxide laser and triamcinolone acetonide
Biological: platelet rich plasma — six sessions of fractional carbon dioxide laser will be done for 10 patients with alopecia areata followed immediately by topical application of autologous platelet rich plasma
  Arms: fractional carbon dioxide laser and platelet rich plasma
Drug: vitamin D solution — six sessions of fractional carbon dioxide laser will be done for 10 patients with alopecia areata followed immediately by topical application of vitamin D solution
  Arms: fractional carbon dioxide laser and vitamin D solution

SUMMARY:
Alopecia areata is a non-scarring hair loss disorder that affects both sexes equally. Incidence of the disease varies for different populations and in different studies, with global incidence ranging from 0.57% to 3.8%.

Etiology of alopecia areata is not completely understood, and the majority of evidence suggests that genetically predisposed individuals, when exposed to an unknown trigger, develop a predominantly autoimmune reaction, leading to acute hair loss. Environmental triggers, including viral or bacterial infections, along with autoimmune disorders, seem to play a major role in the development of alopecia areata.

DETAILED DESCRIPTION:
The onset and progression of alopecia areata are unpredictable. Significant variations in the clinical presentation of alopecia areata have been observed, ranging from small, well-circumscribed patches of hair loss to a complete absence of body and scalp hair.

Although many patients improve spontaneously or respond to standard therapy, treatment can be quite challenging in those with more severe and refractory disease.

Recent advances in the understanding of alopecia areata pathophysiology hold promise for better treatments in the future.

Corticosteroids either topical or intralesional are the most popular drugs for the treatment of this disease. Other therapies like topical minoxidil, anthralin, immunotherapy, systemic corticosteroids, cyclosporine and Psoralen with Ultraviolet-A Light therapy are also commonly used with varying success.

Various lasers have been suggested in recent studies to treat alopecia areata . The effect of 308-nm excimer laser was the most studied, while others, including neodymium-doped yttrium aluminum garnet, erbium:glass laser, fractional carbon dioxide laser, and low-level laser therapy, have also been assessed.

Despite the nascent state of research on lasers as a treatment option for alopecia areata , there have been a great deal of promising results. It is possible for lasers to become the mainstay treatment option of alopecia areata .

It was suggested that ablative fractional lasers may exert its effect through: induction of moderate inflammation to promote anagen entry and creation of channel pathways for topically applied medications they grant access to dermal structures such as hair follicles and cutaneous vasculature. Also, creation of a wound by the ablative fractional laser may stimulate stem cell populations to produce a hair shaft and progress through all stages of the hair follicle cycle.

Majid et al, investigated the efficacy and safety of the combination of fractional carbon dioxide followed by topical triamcinolone acetonide application in ten patients with resistant alopecia areata. Only eight patients completed the study. Seven of them had complete recovery of the treated area. One patient however did not show good response. No significant adverse effects were noted in any of the patients.

The role of platelet rich plasma in promoting hair survival and growth has been demonstrated both in vitro and in vivo. The activation of platelet α granules releases numerous growth factors, including transforming growth factor , platelet derived growth factor, vascular endothelial growth factor, epidermal growth factor, insulin-like growth factor, and interleukin-1. It is proposed that these growth factors may act on stem cells in the bulge area of the follicles, stimulating the development of new follicles and promoting neovascularization. platelet rich plasma has been found to benefit in hair growth in alopecia areata. Intralesional injections of platelet rich plasma were found to increase hair regrowth significantly compared with triamcinolone acetonide or placebo.

Vitamin D 1, 25-dihydroxycholecalciferol [1, 25(OH)/2 D3] is the biologic active form of the vitamin D3. Vitamin D has a multitude of biologic effects interacting with the innate and adaptive immune system, mainly leading to its downregulation. It regulates the differentiation of B cells, T cells, dendritic cells, and the expression of Toll-like receptors. There is growing evidence that vitamin D may help in several autoimmune diseases like multiple sclerosis and type I diabetes mellitus, lupus, and rheumatoid arthritis.

The relation between vitamin D levels and the development of alopecia areata and whether vitamin D supplementation helps in the treatment of alopecia areata represent an attractive area of research. Recent studies suggest that there is deficiency of serum vitamin D and reduced vitamin D receptor expression in the affected hair follicles in alopecia areata patients, the results of which may prove that vitamin D is a safe and helpful choice in alopecia areata treatment.

To the best our knowledge no previous research studied the effect of vitamin D solution in treatment of alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* patients with refractory alopecia areata above 10 years old

Exclusion Criteria:

* Alopecia totalis or alopecia universalis.
* Patients with alopecia other than alopecia areata.
* Patients younger than 10 years.
* Pregnant and lactating females.
* Patients with history of hypertrophic scars or keloid formation.
* Patients with active infection at the site of the lesion.
* Patients with blood disorders and platelet abnormalities and chronic liver disease.
* Patients using anticoagulation therapy and antiplatelet agents.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
response rate | 3 months after last session
  hair regrowth in each group in response to treatment (hair density ) expressed in follicles/ cm2

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Ghazally, MS, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Aksu Cerman A, Sarikaya Solak S, Kivanc Altunay I. Vitamin D deficiency in alopecia areata. Br J Dermatol. 2014 Jun;170(6):1299-304. doi: 10.1111/bjd.12980. PMID 24655364
- [Background] Alkhalifah A, Alsantali A, Wang E, McElwee KJ, Shapiro J. Alopecia areata update: part II. Treatment. J Am Acad Dermatol. 2010 Feb;62(2):191-202, quiz 203-4. doi: 10.1016/j.jaad.2009.10.031. PMID 20115946
- [Background] Huang Y, Zhuo F, Li L. Enhancing hair growth in male androgenetic alopecia by a combination of fractional CO2 laser therapy and hair growth factors. Lasers Med Sci. 2017 Nov;32(8):1711-1718. doi: 10.1007/s10103-017-2232-8. Epub 2017 May 21. PMID 28528395
- [Background] Issa MC, Pires M, Silveira P, Xavier de Brito E, Sasajima C. Transepidermal drug delivery: a new treatment option for areata alopecia? J Cosmet Laser Ther. 2015 Feb;17(1):37-40. doi: 10.3109/14764172.2014.967778. Epub 2014 Oct 16. PMID 25260052